CLINICAL TRIAL: NCT04546867
Title: Sonographic Based Visualization Instead of X-ray of Pancreatic Stents Placed to Prenvent Post-ERCP Pancreatitis.
Brief Title: Establishing a Sonographic Based Algorithm to Verify Pancreatic Stent Position Placed to Prevent Post-ERCP Pancreatitis Before Endoscopic Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Georg Dultz, Principal Investigator, Johann Wolfgang Goethe University Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: FRA-UNI-PANCSTENT-2020
Record Dates: First submitted 2020-08-30; First posted 2020-09-14 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2022-08

CONDITIONS: Post-ERCP Acute Pancreatitis; Pancreatic Stent; Ultrasound; X-rays
Keywords: Post-ERCP Acute Pancreatitis; Pancreatic Stent; Ultrasound; X-rays; Endoscopy; Esophagogastroduodenoscopy

STUDY DESIGN:
Intervention Model Description: The participants will start with a diagnostic ultrasound to visualize a pancreatic stent. If a stent is being displayed in the pancreatic duct. The participants will undergo endoscopy for removal of the pancreatic stent. Otherwise, x-ray will be performed to confirm the sonographic diagnosis. Stents, that are visulized in the duct by x-ray will than be removed. If sonography and x-ray confirm a spontanous dislodgement of the pancreatic stent, no further investigation will be performed.
Masking Description: Neither the investigator nor the patient will know before the sonographic approach, if the pancreatic stent is still in place. The diagnosis will be confirmed either by endoscopic findings or by x-ray depending on sonographic diagnosis and further algorithm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sonography arm (Other): Sonography is being performed by expericenced investigators to visualize a pancreatic stent in the pancreatic duct. If the stent is being visualized, an endoscopy will be performed to remove the stent. Otherwise, x-ray will be needed to confirm the sonographic finding of a dislodged pancreatic stent with no further need of intervention. If x-ray finds a pancreatic stent in situ opposingly to ultrasound, an endoscopy will be performed to confirm the stents position and eventually remove it.
  Interventions: Diagnostic Test: Sonographic based visualization of a pancreatic stent

INTERVENTIONS:
Diagnostic Test: Sonographic based visualization of a pancreatic stent — As described above. All patients start with an ultasound-based approach to visualize pancreatic stents position. Depending on the findings, x-ray will be performed if no stent is visualized in the pancreatic duct or an esophagogastroduodenoscopy will be performed to remove the pancreatic stent and confirm sonographic findings if the pancreatic stent is displayed in situ.

SUMMARY:
The present study is a prospective, single-center study. A total of 88 patients, who had placed a pancreatic stent for preventing post-ERCP pancreatitis, will be included in the study. Aim of the study is to establish a new algorithm based on a sonographic approach to remove the placed pancreatic stents. Another aim is to compare high-end sonographic devices with devices of medium price scale one's used on the ward.

On the day of removal of the pancreatic stent, all patients receive a sonography by an experienced investigator on the ward and by another, uninformed investigator with a high-end device. If a pancreatic stent is visualized in the pancreatic duct, the patient will have an esophagogastroduodenoscopy to remove the pancreatic stent. If sonography cannot find a pancreatic stent in the pancreatic duct an x-ray will be performed as suggested by the European and international guidelines. If the pancreatic stent spontaneously dislocated into the small bowel tract according to x-ray, no further investigation will be performed. If a stent is visulized in situ by x-ray, it will be removed by endoscopyl.

Statistical analysis will be done in cooperation with the statistical biomedical institute oft he university hospital in Frankfurt.

ELIGIBILITY:
Inclusion Criteria:

* placement of prophylactic pancreatic stent to prevent post-ERCP-pancreatitis
* age of at least 18 years
* written informed consent

Exclusion Criteria:

* diseases that prevent sonography, x-ray or esophagogastroduodenoscopy
* no given consent
* other indication for pancreatic stenting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Confirmation of a new algorithm to remove a prophylactic pancreatic stent placed to prevent post-ERCP pancreatitis by using sonography as first approach and compare the findings statistically in a pivot table to x-ray and endoscopy. | The entire procedure will take place within one hour.
  A new algorithm is supposed to be tested that starts with a sonography to display a pancreatic stent. If the pancreatic stent can be visualized in the pancreatic duct, an esophagogastroduodenoscopy will be performed directly to remove the stent. If the stent cannot be displayed by sonography, x-ray will be performed as commonly suggested by the European and international guidelines.
  Therefore, the main goal of the study is to implement sonography before further diagnostic modalities to confirm prophylactic pancreatic stents position in the pancreatic duct.

SECONDARY OUTCOMES:
Comparison of the findings of high-end sonographic devices and the findings of medium prize sonographic devices used on the ward by using a pivot table. | Both will take place within 30 minutes.
  There will be performed two different ultrasounds to confirm stents position by two different experienced investigators. The results will be compared to the results of x-ray and/or endoscopy to evaluate the quality of high end to medium prize sonographic devices.
Univariate analysis of the baseline characteristics compared to the results of sonographic findings to evaluate risk factors of false sonographic findings by using a Case report form to collect the data. | The entire procedure will take place within one hour.
  Baseline characteristics will be compared to the false-positive and false-negative results of sonography compared to the gold standard (x-ray/endoscopy)

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum der J. W. Goethe-Universität, Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Denzer U, Beilenhoff U, Eickhoff A, Faiss S, Huttl P, In der Smitten S, Jakobs R, Jenssen C, Keuchel M, Langer F, Lerch MM, Lynen Jansen P, May A, Menningen R, Moog G, Rosch T, Rosien U, Vowinkel T, Wehrmann T, Weickert U; Deutsche Gesellschaft fur Gastroenterologie, Verdauungs- und Stoffwechselkrankheiten. [S2k guideline: quality requirements for gastrointestinal endoscopy, AWMF registry no. 021-022]. Z Gastroenterol. 2015 Dec;53(12):E1-227. doi: 10.1055/s-0041-109598. Epub 2016 Jan 19. No abstract available. German. PMID 26783975
- [Background] Tryliskyy Y, Bryce GJ. Post-ERCP pancreatitis: Pathophysiology, early identification and risk stratification. Adv Clin Exp Med. 2018 Jan;27(1):149-154. doi: 10.17219/acem/66773. PMID 29521055
- [Background] Cheon YK, Cho KB, Watkins JL, McHenry L, Fogel EL, Sherman S, Lehman GA. Frequency and severity of post-ERCP pancreatitis correlated with extent of pancreatic ductal opacification. Gastrointest Endosc. 2007 Mar;65(3):385-93. doi: 10.1016/j.gie.2006.10.021. PMID 17321236
- [Background] Andriulli A, Loperfido S, Napolitano G, Niro G, Valvano MR, Spirito F, Pilotto A, Forlano R. Incidence rates of post-ERCP complications: a systematic survey of prospective studies. Am J Gastroenterol. 2007 Aug;102(8):1781-8. doi: 10.1111/j.1572-0241.2007.01279.x. Epub 2007 May 17. PMID 17509029
- [Background] Dumonceau JM, Kapral C, Aabakken L, Papanikolaou IS, Tringali A, Vanbiervliet G, Beyna T, Dinis-Ribeiro M, Hritz I, Mariani A, Paspatis G, Radaelli F, Lakhtakia S, Veitch AM, van Hooft JE. ERCP-related adverse events: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2020 Feb;52(2):127-149. doi: 10.1055/a-1075-4080. Epub 2019 Dec 20. PMID 31863440
- [Background] Fan JH, Qian JB, Wang YM, Shi RH, Zhao CJ. Updated meta-analysis of pancreatic stent placement in preventing post-endoscopic retrograde cholangiopancreatography pancreatitis. World J Gastroenterol. 2015 Jun 28;21(24):7577-83. doi: 10.3748/wjg.v21.i24.7577. PMID 26140006
- [Background] Loloi J, Lipkin JS, Gagliardi EM, Levenick JM. Assessing spontaneous passage of prophylactic pancreatic duct stents by X-ray: is a radiology report adequate? Ther Adv Gastrointest Endosc. 2019 Jul 16;12:2631774519862895. doi: 10.1177/2631774519862895. eCollection 2019 Jan-Dec. PMID 31360920
- [Background] Sieg A, Hachmoeller-Eisenbach U, Eisenbach T. Prospective evaluation of complications in outpatient GI endoscopy: a survey among German gastroenterologists. Gastrointest Endosc. 2001 May;53(6):620-7. doi: 10.1067/mge.2001.114422. PMID 11323588
- [Background] ASGE Standards of Practice Committee; Ben-Menachem T, Decker GA, Early DS, Evans J, Fanelli RD, Fisher DA, Fisher L, Fukami N, Hwang JH, Ikenberry SO, Jain R, Jue TL, Khan KM, Krinsky ML, Malpas PM, Maple JT, Sharaf RN, Dominitz JA, Cash BD. Adverse events of upper GI endoscopy. Gastrointest Endosc. 2012 Oct;76(4):707-18. doi: 10.1016/j.gie.2012.03.252. No abstract available. PMID 22985638